CLINICAL TRIAL: NCT02255045
Title: Evaluation of the Effect of a Vaginal Ring With Meloxicam on Primary Dysmenorrhea in Women of Childbearing Age
Brief Title: Assessment of a Vaginal Ring With Meloxicam in the Treatment of Dysmenorrhea
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Laboratorios Andromaco S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AVM002
Record Dates: First submitted 2014-09-22; First posted 2014-10-02 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Meloxicam; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose 1 of meloxicam in vaginal ring (Experimental): 2.4 g of meloxicam in a vaginal ring
  Interventions: Drug: Meloxicam; Drug: Placebo Oral
- Dose 2 of meloxicam in vaginal ring (Experimental): 3.0 g of meloxicam in a vaginal ring
  Interventions: Drug: Meloxicam; Drug: Placebo Oral
- Oral non-steroidal anti-inflammatory drug (Active Comparator): Diclofenac potassium
  Interventions: Drug: Diclofenac Potassium; Drug: Placebo Vaginal
- Placebo vaginal ring and oral pill (Placebo Comparator): Placebo vaginal ring and placebo oral pill
  Interventions: Drug: Placebo Oral; Drug: Placebo Vaginal

INTERVENTIONS:
Drug: Meloxicam — 1 Meloxicam Vaginal Ring (MVR) for 4-6 days
  Arms: Dose 1 of meloxicam in vaginal ring; Dose 2 of meloxicam in vaginal ring
Drug: Diclofenac Potassium — 1 tablet 50 mg diclofenac every 12 hours for 4-6 days
  Arms: Oral non-steroidal anti-inflammatory drug
Drug: Placebo Oral — 1 placebo tablet every 12 hours for 4-6 days
  Arms: Dose 1 of meloxicam in vaginal ring; Dose 2 of meloxicam in vaginal ring; Placebo vaginal ring and oral pill
Drug: Placebo Vaginal — 1 placebo vaginal ring for 4-6 days
  Arms: Oral non-steroidal anti-inflammatory drug; Placebo vaginal ring and oral pill

SUMMARY:
The investigators propose that the sustained administration of a vaginal ring would have a better response with respect to pain and a better safety profile than the oral administration of a non-steroidal anti-inflammatory drug.

To assess the relief of the symptoms associated with dysmenorrhea, a specific survey was elaborated that also includes a Visual Analog Scale (VAS) to objectify and measure dysmenorrhea as is the case with McGill's Pain Questionnaire (MPQ).

ELIGIBILITY:
Inclusion Criteria:

* Regular menstrual cycles on previous 3 months (24-35 days),
* Primary dysmenorrhea on 3 previous months,
* With tubal ligation or users of condom for contraception,
* Hemoglobin of at least 11 g/dl,
* Safety blood analysis in normal levels

Exclusion Criteria:

* Secondary dysmenorrhea,
* Users of hormonal contraceptives (2 months prior to the study) or intrauterine devices (IUDs) (1 month prior the study).
* Allergy to any anti-inflammatory drug including meloxicam or diclofenac.
* Allergy to silicon.
* Pregnant or in lactation.
* Women with untreated or decompensated endocrine disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2014-06-27 (Actual); Primary Completion 2016-02-21 (Actual); Study Completion 2016-03-16 (Actual)

PRIMARY OUTCOMES:
Efficacy: Percentage of primary dysmenorrhea reduction | 5 months
  Change in primary dysmenorrhea using the VAS (0 = pain-free, 10 = maximum pain intensity) for the vaginal ring with meloxicam used during the perimenstrual period compared with a placebo ring.

SECONDARY OUTCOMES:
Minimum effective dose of meloxicam | 5 months
  Determine the minimum effective dose of the vaginal ring with meloxicam in primary dysmenorrhea using a survey. This survey includes a VAS (0 = pain-free, 10 = maximum pain intensity) to evaluate pain intensity, questions about the pain type (superficial, deep), pain location (diffuse, localized), pain duration (for a moment, intermittent, constant), location in the abdominal or back region (yes/no), and the presence of breast pain, thigh pain, mood changes, mastalgia, gastrointestinal disorders, abdominal distension, headache, dizziness, or acne (all with yes/no responses). Furthermore, the survey includes quality of life assessments (effects on routine activity, on work activity and/or housework, social and recreational activities, family and/or interpersonal relationships, state of mind, and sleep quality: 0 = no negative effect, 10 = maximum negative effect).
Efficacy: Comparison of meloxicam vaginal ring and oral diclofenac | 5 months
  Compare the effect of a vaginal ring with meloxicam versus the oral administration of a non-steroidal anti-inflammatory drug commonly used for primary dysmenorrhea during one menstrual cycle, using a survey. This survey includes a VAS (0 = pain-free, 10 = maximum pain intensity) to evaluate pain intensity, questions about the pain type (superficial, deep), pain location (diffuse, localized), pain duration (for a moment, intermittent, constant), location in the abdominal or back region (yes/no), and the presence of breast pain, thigh pain, mood changes, mastalgia, gastrointestinal disorders, abdominal distension, headache, dizziness, or acne (all with yes/no responses). Furthermore, the survey includes quality of life assessments (effects on routine activity, on work activity and/or housework, social and recreational activities, family and/or interpersonal relationships, state of mind, and sleep quality: 0 = no negative effect, 10 = maximum negative effect).

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (1):
- Instituto Chileno de Medicina Reproductiva (ICMER), Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marjoribanks J, Proctor M, Farquhar C, Derks RS. Nonsteroidal anti-inflammatory drugs for dysmenorrhoea. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD001751. doi: 10.1002/14651858.CD001751.pub2. PMID 20091521
- [Background] Harel Z. Cyclooxygenase-2 specific inhibitors in the treatment of dysmenorrhea. J Pediatr Adolesc Gynecol. 2004 Apr;17(2):75-9. doi: 10.1016/j.jpag.2004.01.002. PMID 15050982
- [Background] de Mello NR, Baracat EC, Tomaz G, Bedone AJ, Camargos A, Barbosa IC, de Souza RN, Rumi DO, Martinez Alcala FO, Velasco JA, Cortes RJ. Double-blind study to evaluate efficacy and safety of meloxicam 7.5 mg and 15 mg versus mefenamic acid 1500 mg in the treatment of primary dysmenorrhea. Acta Obstet Gynecol Scand. 2004 Jul;83(7):667-73. doi: 10.1111/j.0001-6349.2004.00433.x. PMID 15225193
- [Background] Chantler I, Mitchell D, Fuller A. The effect of three cyclo-oxygenase inhibitors on intensity of primary dysmenorrheic pain. Clin J Pain. 2008 Jan;24(1):39-44. doi: 10.1097/AJP.0b013e318156dafc. PMID 18180635